CLINICAL TRIAL: NCT03551951
Title: Tumor Cell and DNA Detection in the Blood, Urine and Bone Marrow of Patients With Solid Cancers and Subjects Undergoing Lung Cancer Screening
Brief Title: Tumor Cell and DNA Detection in the Blood, Urine, and Bone Marrow
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Harry S. Truman Memorial Veterans' Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jussuf Kaifi, Assistant Professor, Chief, Thoracic Surgery, University of Missouri-Columbia
Other Study IDs: 2004401-VA
Record Dates: First submitted 2018-05-23; First posted 2018-06-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Hepatocellular Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, lymphocyte DNA, urine, bone marrow, cancer tissue, healthy tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients having surgery: Cancer patients undergoing surgery will have test for circulating tumor cells, DNA alterations
  Interventions: Diagnostic Test: Test for circulating tumor cells, DNA alterations
- Patients not having surgery: Cancer patients not undergoing surgery (but potentially other treatments) will have test for circulating tumor cells, DNA alterations.
  Lung cancer screening subjects
  Interventions: Diagnostic Test: Test for circulating tumor cells, DNA alterations
- Healthy subjects: Healthy control subjects will have test for circulating tumor cells, DNA alterations
  Interventions: Diagnostic Test: Test for circulating tumor cells, DNA alterations

INTERVENTIONS:
Diagnostic Test: Test for circulating tumor cells, DNA alterations

SUMMARY:
Patients with resectable solid primary cancers and even limited number of metastases are potentially curable. However, most patients develop recurrences despite surgery. Also, early detection of lung cancer with low dose CT screening may cure patients at an early stage. Circulating and disseminated tumor cell (CTC/DTC) and circulating cell-free (cf) DNA isolation from the blood, urine and bone marrow will increase understanding of cancer spread and advance knowledge to develop individualized therapies and improve screening.

DETAILED DESCRIPTION:
Background: Patients with resectable solid primary cancers and even limited number of metastases are potentially curable. However, most patients develop recurrences despite surgery. Circulating and disseminated tumor cell (CTC/DTC) and circulating cell-free (cf) DNA isolation from the blood, urine and bone marrow will increase understanding of cancer spread and advance knowledge to develop individualized therapies. These liquid biomarkers might also be suitable for screening purposes and early detection of in high risk subjects for lung cancer.

Hypothesis and Rationale: CTCs/DTCs and cfDNA isolated from the blood, urine and bone marrow undergo pheno- and/or genotype changes. CTCs/DTCs have potential for dissemination and tumor growth in vivo. Investigating the biology of liquid biomarkers in the blood, urine and bone marrow will significantly increase understanding of cancer biology of early and advanced stages.

Specific Aims: CTCs/DTCs and cfDNA will be quantified and characterized for genetic alterations and expression of key signaling/proliferation biomarkers and grow in vivo in nude mice.

Study Design: 100 cancer patients will be recruited for CTC/DTC/cfDNA isolation from the blood, urine and bone marrow with innovative techniques. Bone marrow will be drawn only perioperatively in cancer patients undergoing anesthesia for surgery. 200 high-risk individuals undergoing lung cancer screening with a low dose CT will also be included for blood and urine collection to test the usefulness of these liquid biomarkers for early detection of lung cancer. In addition, 20 individuals with benign disease will also be included as controls. CTCs/DTCs, cfDNA and cancer tissue pheno- and/or genotype analysis will be performed with different innovative techniques. Furthermore, CTCs/DTCs will be enriched, cultured and characterized. Tumor growth potential will be studied in nude mice.

Relevance: This study addresses fundamental aspects of cancer disease being the cause of death in 1 out of 4 persons in the US. Innovative CTCs/DTCs characterization can shed light on the tumor biology, and identify therapy targets. Results of this study can be fundamentally important to understanding cancer spread and development of personalized therapies, and improve early detection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years.
* Subjects of all genders and ethnicities.
* Subjects with the diagnosis of a solid cancer (n=100) of all stages will be included (lung, esophageal, stomach, bile duct/pancreas, colorectal, melanoma, sarcoma).
* Ten patients with no present suspicion and no previous history of any cancer (except basal cell cancer of the skin) that undergo surgeries for other benign indications will serve as controls (n=10).
* In patients undergoing surgery for cancer the histopathology should preferably be pathologically proven by a previous or novel biopsy. Yet, patients with a high cancer suspicion by radiology and clinical picture that undergo cancer surgery will not be excluded. No additional biopsies, testing or interventions will be performed for the purpose of this study if the medical treatment will not require it.
* Subjects must be capable of giving informed consent.
* Lung cancer screening eligibility criteria (n=100): 55-80 years old, >30 pack years smoking history, and current smoker or have quit within the last 15 years)

Exclusion Criteria:

* Pregnant women.
* Subjects with the concurrent diagnosis of an active secondary (synchronous) malignancy besides basal cell carcinoma of the skin will be excluded, if there is evidence of disease burden or if the patient is currently being treated with chemotherapy.
* Subjects with a hemoglobin of <8g/dl in the morning of the procedure will be excluded.
* In subjects who require intraoperative transfusions of >4 units of red packed blood cells (RPBCs), no further blood will be drawn for CTC/DTC/cfDNA analysis during surgery or on postoperative day 1.
* In patients with coagulation disorders that could lead to significant bleeding (such as hemophilia, significant thrombocytopenia) requiring prophylactic administration of coagulative products, no bone marrow aspiration will be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with the diagnosis of a solid cancer of all stages will be included (lung, esophageal, stomach, bile duct/pancreas, colorectal, melanoma, sarcoma).
  Lung cancer screening subjects will also be included (as defined above)
  Total recruitment: 320
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of CTC/DTC in blood | At baseline
  Quantify the number of CTC and DTC in urine
Number of CTC/DTC in urine | At baseline
  Quantify the number of CTC and DTC in urine
Number of CTC/DTC in bone marrow | At baseline
  Quantify the number of CTC and DTC in bone marrow
Quantity of cfDNA in blood | At baseline
  Quantify the amount of cfDNA in blood
Quantity of cfDNA in urine | At baseline
  Quantify the amount of cfDNA in urine
Quantity of cfDNA in bone marrow | At baseline
  Quantify the amount of cfDNA in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Jussuf T Kaifi, MD, Principal Investigator — University of Missouri Health Care
Locations (1):
- Harry S Truman Veterans Memorial Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
no data will be shared